CLINICAL TRIAL: NCT04314245
Title: Diagnostic Evaluation of Urine DNA Methylation/Somatic Mutation Profiling for the Detection of Urothelial Carcinoma
Status: Completed | Type: Observational
Sponsor: AnchorDx Medical Co., Ltd. (Industry)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); West China Hospital (Other); RenJi Hospital (Other); Tongji Hospital (Other); Peking University People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Southern Medical University, China (Other); Nanfang Hospital, Southern Medical University (Other); Sichuan Cancer Hospital and Research Institute (Other); Affiliated Hospital & Clinical Medical College of Chengdu University (Unknown)
Responsible Party: Sponsor
Other Study IDs: AnchorDx-BC004
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: Bladder Cancer; Urine; DNA methylation; Somatic mutation
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Urothelial carcinoma group: Subjects who diagnosed with incident or recurrent urothelial carcinoma (including bladder/ureter/renal pelvis) by surgical pathology.
  Interventions: Other: Active Comparator: Pathology; Other: Genetic test: AnchorDx's urine DNA methylation/somatic mutation profiling assay
- interference group: Subjects who diagnosed with incident or recurrent bladder cancer other than urothelial carcinoma (including bladder squamous cell carcinoma/bladder adenocarcinoma/other bladder-related cancers/prostate cancer/rectal cancer) by surgical pathology.
  Interventions: Other: Active Comparator: Pathology; Other: Genetic test: AnchorDx's urine DNA methylation/somatic mutation profiling assay
- Control group: Subjects who clinically diagnosed with benign disease of the urinary system, such as Urinary calculi, urinary tract infection (except urinary tuberculosis), benign prostatic hyperplasia, glandular cystitis.
  Interventions: Other: Active Comparator: Clinical Diagnosis; Other: Genetic test: AnchorDx's urine DNA methylation/somatic mutation profiling assay
- Healthy volunteers group: Volunteers who have a normal routine urine test / ultrasound examination of the urinary system and do not carry suspected tumors of other organs.
  Interventions: Other: Active Comparator: Clinical diagnosis; Other: Genetic test: AnchorDx's urine DNA methylation/somatic mutation profiling assay

INTERVENTIONS:
Other: Active Comparator: Pathology — Routine treatment for bladder cancer, and surgical pathology for confirmation of patients with urothelial carcinoma.
  Groups: Urothelial carcinoma group; interference group
Other: Active Comparator: Clinical Diagnosis — Routine clinical diagnosis and treatment of benign disease of the urinary system
  Groups: Control group
Other: Active Comparator: Clinical diagnosis — Routine urine test and imaging diagnostic techniques, such as B-ultrasound.
  Groups: Healthy volunteers group
Other: Genetic test: AnchorDx's urine DNA methylation/somatic mutation profiling assay — A urine-based assay for the detection of urothelial carcinoma using urine DNA methylation/somatic mutation profiling analysis.

SUMMARY:
Clinical trial to evaluate the performance characteristics(sensitivity and specificity) of AnchorDx's urine DNA methylation/somatic mutation profiling assay for detecting urothelial carcinoma compared to pathology in patients.

DETAILED DESCRIPTION:
This is a prospective study that involves 11 centers in China and 1200 participants. The assay analyzes the DNA methylation/somatic mutation profiles of bladder cancer-specific biomarkers non-invasively using urine specimens collected before invasive diagnosis/treatment. The performance characteristics(sensitivity and specificity) of the assay for detection of urothelial carcinoma is evaluated in comparison to pathology or cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Urothelial carcinoma group:

   * Any male or female patient aged 18 or older.
   * Able to provide urine specimen (100ml for both first void and non-first-void urine) before treatments.
   * Diagnosed with incident or recurrent urothelial carcinoma (including bladder/ureter/renal pelvis) by surgery.
2. interference group:

   * Any male or female patient aged 18 or older.
   * Able to provide urine specimen (100ml for both first void and non-first-void urine) before treatments.
   * Diagnosed with incident or recurrent bladder cancer other than urothelial carcinoma (including bladder squamous cell carcinoma/bladder adenocarcinoma/other bladder-related cancers/prostate cancer/rectal cancer) by surgery.
3. Control group:

   * Any male or female patient aged 18 or older.
   * Able to provide urine specimen (100ml for both first void and non-first-void urine) before treatments.
   * Diagnosed with urinary disease such as Urinary calculi, urinary tract infection (except urinary tuberculosis), benign prostatic hyperplasia, glandular cystitis. All enrollee are able to provide legally effective informed consent.
4. Healthy volunteers group:

   * Any male or female patient aged 18 or older.
   * Able to provide urine specimen (100ml for both first void and non-first-void urine) before physical examination.

exclusion criteria:

1. Urothelial carcinoma/Interference group/Control group

   * Has had diagnosed with other cancers.
   * Patients diagnosed with non-urological cancer.
   * Failed to provide a written informed consent.
2. Healthy volunteers group:

   * Volunteers with abnormal test results of urine analysis or urological ultrasound test.
   * Volunteers sceptical of cancers from non-urological origin in a normal results of urine analysis or urological ultrasound.
   * Failed to provide legally effective informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects consisted of four types : 1) Patients with urothelial carcinoma; 2) Patients with the other bladder cancer (including bladder squamous cell carcinoma/bladder adenocarcinoma/other bladder-related cancers/prostate cancer/rectal cancer); 3) Patients with benign disease of the urinary system, such as Urinary calculi, urinary tract infection (except urinary tuberculosis), benign prostatic hyperplasia, glandular cystitis; 4) Healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 1170 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Performance for the detection of urothelial carcinoma | 1 Years
  The efficacy of the urine DNA methylation/somatic mutation profiling assay for the detection of urothelial carcinoma comparing with pathologic diagnosis, including sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), positive likelihood ratio (+LR), negative likelihood ratio (-LR) and accuracy.

SECONDARY OUTCOMES:
Sensitivity and Specificity in different pathological stages and histologic grades of urothelial carcinoma | 1 Years
  Sensitivity and specificity of urine DNA methylation/somatic mutation profiling assay in different pathological stages and histologic grades of urothelial carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Jian HUANG, MD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No